CLINICAL TRIAL: NCT05772572
Title: Functional Disorders in the MoyaMoya Disease of Children, Adolescents and Young Adults: Place of Anxiety, Depression, Attachment of the Child and Parents, and Representations of Illness and Child Surgery
Brief Title: Functional Disorders Moya Moya Young Patients
Acronym: TFMoya : ADAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220991; 2021-A02555-36 (Other: IDRCB Number)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Moyamoya Disease
Keywords: Moyamoya Disease; Anxiety; Depression; Parent-child attachment; Psychological representations of illness and surgery
MeSH Terms: conditions — Moyamoya Disease; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Children aged 7 to 17 inclusive, and young adults operated (or re-operated) for a Moya Moya in the previous 7 years and followed at the Necker-Enfants Malades hospital, and their parents.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires are completed only once and assess:
  * recorded questions about the disease and the operation for the parents and the patient, human figure drawing test and drawing of the operation for the patient
  * psychiatric questionnaires for parents and patients on anxiety and depression
  * behavior questionnaires for the parents and the patient: assessment of attachment
  * questionnaires for the parents and the patient concerning the family context, the quality of life

SUMMARY:
Moya Moya disease is a rare condition of the vessels that supply blood to the brain. It normally occurs without apparent cause. In both children and adults, the disease is mainly manifested by strokes. Diagnosis is made on MRI and cerebral angiography. There is no treatment that can prevent the arteries in the brain from narrowing.

Surgical treatment may be a priority, especially in the early forms of the disease. Functional, painful disorders, in particular headaches, may persist after neurosurgical intervention, without any clear predictive factor being found. Otherwise there is a disjunction between the objectification of sequelae on MRI and painful complaints, sometimes a dissociation between the improvement of the objective parameters of perfusion and imaging, and functional somatic complaints.

The study focuses on improving knowledge of post-operative functional disorders in Moya Moya disease in children and adolescents, in order to propose interventions based on this knowledge and making it possible to reduce both functional complaints and depression, the anxiety which accompanies them, to decrease the impact on the quality of life and parental wandering in the installation of adapted accompaniments. For this, a half-day consultation will be intended in order to carry out questionnaires and standardized tests, the results of which will be reported and compared to known rates in the general population and the population of children with chronic diseases.

DETAILED DESCRIPTION:
Moya Moya disease is a rare condition of the vessels that supply blood to the brain. It normally occurs without apparent cause. In both children and adults, the disease is mainly manifested by strokes. Diagnosis is made on MRI and cerebral angiography. There is no treatment that can prevent the arteries in the brain from narrowing.

Surgical treatment can be considered, especially in the early forms of the disease. Several surgical techniques are used to divert the vessels, including multiple craniotomies, which consists of making several small holes in the cranium so as to pass vessels from the scalp so that they develop towards the poorly irrigated areas of the brain.

Functional, painful disorders, in particular headaches, can persist after neurosurgical intervention, without any clear predictive factor being found. 57% of patients under 17 with Moya Moya disease have persistent functional disorders in without correlation to any of the characteristics of the disease, nor to its surgical treatment. There is a disjunction between the objectification of sequelae on MRI and painful complaints, sometimes a dissociation between the improvement of the objective parameters of perfusion and imaging, and functional somatic complaints. Interviews with families experienced that psychological phenomena may play an important role in postoperative pain and functional complaints: child and parent anxiety, depression, and family functioning and attachment, child cognitive functioning.

Functional complaints and postoperative pain are therefore frequent in children and adolescents with Moya Moya, but poorly documented. The difficulty is to be able to disentangle the pain linked to organic factors such as a recurrence of a vascular accident, and those linked to psychological factors, as they have been described in the disease. The important thing is to be able to avoid or reduce paraclinical explorations in the face of the resurgence of painful complaints; the challenge is to defuse the vicious interactive circle between painful complaints, anxiety-provoking explorations, reinforcing stress and possible increase complaints. Identifying the psychological factors would make it possible to better support functional complaints.

The study focuses on improving knowledge of post-operative functional disorders in Moya Moya disease in children and adolescents, in order to propose interventions based on this knowledge and making it possible to reduce both functional complaints and depression, the anxiety which accompanies them, to decrease the impact on the quality of life and parental wandering in the installation of adapted accompaniments. For this, a half-day consultation will be intended in order to carry out questionnaires and standardized tests, the results of which will be reported and compared to known rates in the general population and the population of children with chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients up to 25 years old and minor patients aged 7 to 17 inclusive and holders of parental authority for minor patients
* Patients operated (or re-operated) for a Moya Moya in the previous 7 years
* Subjects without intellectual disabilities
* Subjects speaking French well enough to answer the questions of the study
* subjects (parent(s) and minor or adult patient) and holders of parental authority informed and who do not object to their participation in the study

Exclusion Criteria:

Cognitive level of the patient incompatible with the administration of the questionnaires and evaluations of the study

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The cohort will be selected from the Necker Hospital cohort (child neurology and neurosurgery services).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
The " State trait anxiety inventory ", STAI forme Y | Day 0
  Study the links between postoperative functional disorders by multiple craniotomies in children and adolescents with Moya Moya disease, and psychological dimensions such as anxiety.
  For teenager, adults patients and parents : The " State trait anxiety inventory ", STAI form Y (revised), a self-questionnaire assessing trait anxiety (usual tendency to be anxious) and state anxiety (anxiety felt at a particular time), has 20 items for assessing trait anxiety and 20 for state anxiety on a 4-point Likert scale, scores range from 20 to 80, with higher scores correlating with greater anxiety.
Revised Children's Manifest Anxiety Scale (RCMAS) | Day 0
  Revised Children's Manifest Anxiety Scale (RCMAS) : self-administered 37-item questionnaire assessing the level and nature of anxiety in children and adolescents aged 9 to 19, not allowing diagnosis of the various anxiety disorders in children. The total anxiety score can range from 0 to 28. The cut-off point for pathological anxiety is more than two standard deviations around the mean (T more than 70).
Children Depression Inventory (CDI) | Day 0
  Study the links between postoperative functional disorders by multiple craniotomies in children and adolescents with Moya Moya disease, and psychological dimensions such as depression.
  CDI Children Depression Inventory : self questionnaire of 27 items which measures the intensity of depression in children and adolescents from 7 to 17 years old. Each item is rated from 0 (normal behavior for age or absent) to 2 (severe). The addition of the items gives a total between 0 and 54. The higher the score, the more severe the depression symptomatology is.
Beck = Depression | Day 0
  Parents and young adult patients : Beck = Depression Multiple-choice questionnaire of 21 items of symptoms and attitudes, used to measure the severity of clinical depression, graded from 0 to 3 by a series of 4 statements (from 0 to 63, higher score correlating with higher severity) reflecting the degree of severity of the symptom.
FMSS= Five minute speech sample, quality of the parent-child relationship | Day 0
  The Five Minute Speech Sample (FMSS) is a method that can be used to measure both expressed emotion and narrative coherence. The FMSS requires parents to speak about their child and their relationship with their child for five minutes. The final coding assesses one of two categories: high Expressed Emotions (H EE), or Low Expressed Emotions (Low EE).
Cards for the evaluation of Attachment and Mentalization in Children (CAME) | Day 0
  Study the links between postoperative functional disorders by multiple craniotomies in children and adolescents with Moya Moya disease, and psychological dimensions such as of attachment of child with parents.
  CAME: Cards for the evaluation of Attachment and Mentalization in Children, from Child Attachment Interview. The final coding assesses 6 principal dimensions of attachment and 8 secondary dimensions in T quantitative scores. The T scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points. Higher scores indicate greater problems. Principal attachment dimensions: Secure (SEC), Insecure-Deactivated (DEAC), Insecure-Hyperactivated (HYP), insecure disorganized (DIS), Mentalized Attachment (MENT-A); the 8 secondary dimensions are: Coherence (COH), Reflective Self (REF-S), Access to Memories (MEM), Mentalization (MENT), Preoccupation/anger (PRE-A), Traumatism (TRAU), Need comfort (COM), Life Difficulties (LIFE-D).
CA-MIR : cards for assessment of parent's attachment | Day 0
  Cards for assessment of parent's attachment. The final coding assesses 3 principal dimensions of attachment and 13 secondary dimensions in T quantitative scores. The standard scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points. Higher scores indicate greater problems.
  Principal attachment dimensions: Secure (SEC), Insecure- Detached (DET), Insecure- Preoccupied (PRE); the 13 secondary dimensions are : Parental Interference (PAR-I), Family concern (FAM-C), Infantilization Grudge (INF-G), Parental support (PAR-S), Family support (FAM-S), Recognition of support (REC-SUP), Parental unavailability (PAR-UN), Family (FAM-D), Rejection Grudge (REJ-G), Parental Trauma (PAR-TR), Memory Blocking (MEM-B), Parental resignation (PAR-RE), Valuation of Hierarchy (HIE-V).
Child Behavior Checklist (CBCL) | Day 0
  The Child Behavior Checklist (CBCL) is a checklist parents complete to detect emotional and behavioural problems in children and adolescents.
  The main scoring for the CBCL is based on statistical groupings of sets of behaviors that typically occur together.
  Coding assesses 8 syndrome scales:withdrawal, somatic complaints, anxious/depressed, social problems, thought problems, attention problems, rule-breaking behaviour, aggressive behaviour, and two higher order factors: internalizing, and externalizing, and a total score.The standard scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points.
  For each syndrome, Internalizing and Externalizing problem scales, and the total score, scores can be interpreted as falling in the normal, borderline, or clinical behavior.
Representations of disease and surgery | Day 0
  Human figure drawing test and drawing of the operation for the patient. Recorded questions about the disease and the operation for the parents and the patient.
  * For the human figure: The Royer grid will allow to define 1) quartiles for the size of the figure according to the age of the child 2) the developmental age for the figure, according to a score varying from 0 to 60.
  * responses will be qualitatively analyzed to determine prevalent themes.
Pediatric Quality of Life Inventory (PedsQL) | Day 0
  The Pediatric Quality of Life Inventory (PedsQL) makes it possible to assess the quality of life in relation to the state of health of healthy children or children suffering from various diseases. The 23 questions, each scoring from 0 (never) to 4 (almost always), relate to 4 different areas: the functional physical (8 items, total from 0 to 32), emotional (5 items, total from 0 to 20), social (5 items, total from 0 to 20), and school (5 items, total from 0 to 20). A total score can be calculated (from 0 to 92).
  4 versions are proposed, according to the age of the child/adolescent/young adult, each scoring in the same way.

SECONDARY OUTCOMES:
Medical and neuropsychological assessment of patients | Day 0
  1. association between medical parameters (history of stroke, number of surgical procedures, hypoperfusion on MR imaging, or cognitive dysfunction) and presence of functional disorders
  2. association between medical parameters (history of stroke, number of surgical procedures, hypoperfusion on MR imaging, or cognitive dysfunction) and anxiety (RCMAS score >70), depression (abnormal Beck score), or functional attachment (abnormal high CAME score)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ouss, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Manoelle Kossorotoff, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No